CLINICAL TRIAL: NCT03580187
Title: Nebulized Morphine in Chest Trauma Patients: A Prospective Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Mahdia (Other)
Responsible Party: Principal Investigator, Majdoub Ali MD, head of anesthesia departement, University Hospital, Mahdia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMCT/1
Record Dates: First submitted 2018-06-14; First posted 2018-07-09 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Blunt Injury of Thorax
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Intervention Model Description: Were included all patients aged 18 years and over, victims of isolated chest trauma, who were admitted to the intensive care unit. We excluded patients with any of the following criteria: not consent, pregnant woman, polytrauma, hemodynamic instability with systolic blood pressure less than 100 mmHg, treatment with morphine during transport or in the emergency room, need for initial ventilatory support, bradypnea (respiratory rate less than 12 cycles per minute), allergy to opiods, initial pain Visual Analog Scale (VAS) ≤ 4. Pain level was assessed by the pain VAS. We collected demographic, epidemiological, initial clinical examination data, explorations, lesions and we monitored the evolution of the VAS and the vital signs. Informed consent was obtained from all patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- morphine + (Other): We performed a first nebulization of 10 mg (1mL) of morphine diluted in 4 mL of normal saline using a nebulizer with an oxygen flow rate of 8 L / min. The quality of analgesia was assessed by VAS at rest and cough after 10 minutes. If ≤ 4, we concluded to a success. If VAS was still> 4, a second nebulization was performed. After 20 minutes, if VAS still higher than 4 we performed a third nebulization. If pain level was ≤ 4, we concluded to a success.
  morphine (+) group: good response to morphine in nebulization after 30 min if VAS > than 4 we conclude to morhine (-)
  Interventions: Drug: Morphine (+)

INTERVENTIONS:
Drug: Morphine (+) — We performed a first nebulization of 10 mg (1mL) of morphine diluted in 4 mL of normal saline using a nebulizer with an oxygen flow rate of 8 L / min. The quality of analgesia was assessed by VAS at rest and cough after 10 minutes. If ≤ 4, we concluded to a success. If VAS was still> 4, a second nebulization was performed. After 20 minutes, if VAS still higher than 4 we performed a third nebulization. If pain level was ≤ 4, we concluded to a success. After 30 minutes, if VAS still> 4, we concluded to a failure of morphine nebulization.
  The patients were divided into two groups:
  morphine (+) group: good response to morphine in nebulization morphine (-) group: failure of morphine in nebulization
  Other Names: morphine (-)

SUMMARY:
This is a prospective study carried out from 2018 to 2020 including patients aged ≥ 18 years, admitted for isolated chest trauma. Each patient received a nebulization of 10 mg morphine. If Visual Analog Score (VAS) assessed after 10 minutes still> 4, nebulization was repeated every 10 minutes until pain relief. At 30 minutes, VAS> 4 means failure.

DETAILED DESCRIPTION:
The aim of this study was to determine the predictive factors of nebulized morphine failure in patients with chest trauma and to establish a score based on these factors to guide the analgesic protocol.

Methods: This is a prospective study carried out from 2018 to 2020 including patients aged ≥ 18 years, admitted for isolated chest trauma. Each patient received a nebulization of 10 mg morphine. If Visual Analog Score (VAS) assessed after 10 minutes still> 4, nebulization was repeated every 10 minutes until pain relief. At 30 minutes, VAS> 4 means failure.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years and over
* victims of isolated chest trauma,
* admitted to the intensive care unit

Exclusion Criteria:

* not consen
* pregnant woman
* polytrauma
* hemodynamic instability with systolic blood pressure less than 100 mmHg,
* treated with morphine during transport or in the emergency room
* need initial ventilatory support, bradypnea (respiratory rate less than 12 cycles per minute)
* allergy to opiods
* initial pain Visual Analog Scale (VAS) ≤ 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
analgesia evaluated with visual scale | 30 minuts
  morphine (+) group: good response to morphine in nebulization morphine (-) group: failure of morphine in nebulization

CONTACTS AND LOCATIONS:
Locations (1):
- Mahdia Hospital, Mahdia, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Attia H, Ben Saad H, Masmoudi K, Bannour I, Ouaz M, Gardabbou K, Majdoub A. Predictive factors of nebulized morphine failure in North-African patients with chest trauma: a prospective pilot study. Expert Rev Respir Med. 2022 Oct;16(10):1085-1092. doi: 10.1080/17476348.2022.2131543. Epub 2022 Oct 5. PMID 36196899